CLINICAL TRIAL: NCT02920268
Title: Just in TIME - Intervention With Dance and Yoga for Girls With Recurrent Abdominal Pain
Acronym: Just in TIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Duberg (Other)
Collaborators: Örebro University, Sweden (Other); Region VÃ¤stmanland (Unknown)
Responsible Party: Sponsor-Investigator, Anna Duberg, PhD, Region Örebro County
Organization: Region Örebro County (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 209695
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Functional Abdominal Pain; IBS
Keywords: dance-intervention; yoga; adolescents; recurrent abdominal pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intervention with dance and yoga sessions, two times a week in 8 months.
  Interventions: Other: Dance and yoga intervention
- Controls (No Intervention): No intervention

INTERVENTIONS:
Other: Dance and yoga intervention
  Arms: Intervention

SUMMARY:
Recurrent abdominal pain affects up to 37% of school-age children, mostly girls. These problems results in decreased quality-of-life, absence from school, lower sleep quality and increased health-care consumption. Long-term effects are lasting pain-symptoms and increased risk for psychiatric illness.

The scientific evidence for interventions towards long-term pain in children is limited and pharmacological treatment is not effective. Cognitive behavioral therapy has shown some effect but is time- and resource consuming. Dance and yoga can enhance positive protective factors through better body awareness and increased self-regulation. Relaxation in yoga also has positive effect on abdominal pain.

The aim of this study is to evaluate the effects of an intervention with dance and yoga for girls, 9 to 13 years old, with recurrent abdominal pain. The participants will be identified through pediatric clinics in Örebro County, primary health care and school health care. They will be randomized to intervention with weekly dance- and yoga class for 8 months or control group with standard treatment. Primary outcome is the fraction of girls in each group who, direct after intervention, has decreased their maximum pain measured by Faces Pain Scale. Secondary outcomes are stress, psychical health, well-being, school and sleep functions, physical activity and health-economy. The study group will be followed up for two years.

Just-in-TIME is an interdisciplinary research group with expertise in interventions for psychosomatic problems in children and adolescents. TIME, which stands for Try, Identify, Move and Enjoy, also characterizes this project, aiming at decreasing recurrent abdominal pain through an intervention with dance and yoga for 9-13 year old girls.

ELIGIBILITY:
Inclusion Criteria:

Girls 9-13 years old as of pediatricians receive or have received the diagnosis functional abdominal pain or IBS according to the ROME III criteria and stating that they have persist symptoms for at least 2 months after completed investigation from pediatricians. Persistent symptoms are measured by pain diary at baseline and means that the girl at least once in the pain diary estimates 4 or higher as measured by the Faces Pain Scale (FPS-R).

Exclusion Criteria:

* Simultaneous celiac disease or inflammatory bowel disease (IBD).
* Difficulties in following verbal instructions such as hearing impaired or mentally retarded.
* Girls who are deemed to have such serious psychological symptoms that other treatment is required. All participants in the study, which estimates over 13 at the Children's Depression Screener (Child-S), will meet a psychologist / psychiatrist to assess whether they can participate in the study or have direct access to the Children and Youth psychiatry.
* Children treated with CBT.

Ages: 9 Years to 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Faces pain scale (FPS-R) | Immediately after the intervention compared to the control group
  Has the perceived abdominal pain decreased by a 8 months long intervention with regular dance and yoga for girls with recurrent abdominal pain, measured immediately after the intervention compared to the control group? The primary outcome is the proportion of girls in each group that have lowered their maximal abdominal pain measured by Faces Pain Scale (FPS-R).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Duberg, PhD, Principal Investigator — University health care research center, Region Örebro county
Locations (1):
- University health care research center, Region Örebro county, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duberg A, Eriksson M, Philipson A. Parent-child agreement in reporting somatic distress, gastrointestinal symptoms, mental health, and general health in girls with functional abdominal pain. Eur J Pediatr. 2025 Nov 22;184(12):780. doi: 10.1007/s00431-025-06640-5. PMID 41273450
- [Derived] Hogstrom S, Eriksson M, Morelius E, Duberg A. "A source of empowerment and well-being": Experiences of a dance and yoga intervention for young girls with functional abdominal pain disorders. Front Pediatr. 2023 Apr 21;11:1040713. doi: 10.3389/fped.2023.1040713. eCollection 2023. PMID 37152307
- [Derived] Philipson A, Duberg A, Hagberg L, Hogstrom S, Lindholm L, Moller M, Ryen L. The Cost-Effectiveness of a Dance and Yoga Intervention for Girls with Functional Abdominal Pain Disorders. Pharmacoecon Open. 2023 Mar;7(2):321-335. doi: 10.1007/s41669-022-00384-w. Epub 2023 Jan 16. PMID 36646863
- [Derived] Hogstrom S, Philipson A, Ekstav L, Eriksson M, Fagerberg UL, Falk E, Moller M, Sandberg E, Sarnblad S, Duberg A. Dance and yoga reduced functional abdominal pain in young girls: A randomized controlled trial. Eur J Pain. 2022 Feb;26(2):336-348. doi: 10.1002/ejp.1862. Epub 2021 Sep 21. PMID 34529293
- [Derived] Philipson A, Sarnblad S, Ekstav L, Eriksson M, Fagerberg UL, Moller M, Morelius E, Duberg A. An Intervention With Dance and Yoga for Girls With Functional Abdominal Pain Disorders (Just in TIME): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Dec 15;9(12):e19748. doi: 10.2196/19748. PMID 33320103